CLINICAL TRIAL: NCT05151640
Title: Prospective Observational Investigation of Possible Correlations Between Change in FVC and Change in Cough or Dyspnea Scores Using the Living With Pulmonary Fibrosis Questionnaire (L-PF) Between Baseline and After Approximately 52 Weeks of Nintedanib Treatment in Patients Suffering From Chronic Fibrosing ILD With a Progressive Phenotype
Brief Title: INCHANGE - Nintedanib for Changes in Cough and Dyspnea in Patients Suffering From Chronic Fibrosing Interstitial Lung Disease With a Progressive Phenotype in Everyday Clinical Practice: a Real-world Evaluation
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0467
Record Dates: First submitted 2021-12-01; First posted 2021-12-09 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nintedanib treatment group
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib

SUMMARY:
The primary objective of this study is to investigate the correlation between changes from baseline to 52 weeks in Forced Vital Capacity (FVC) [% pred.] and changes from baseline to 52 weeks in dyspnea score [points] or cough score [points] as measured with the living with pulmonary fibrosis (L-PF) questionnaire over 52 weeks of nintedanib treatment in patients suffering from chronic fibrosing Interstitial lung disease (ILD) with a progressive phenotype (excluding idiopathic pulmonary fibrosis (IPF)).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years at Visit 1
* Subjects must be contractually capable and mentally able to understand and follow the instructions of the study personnel
* Physician's diagnosis of chronic fibrosing Interstitial lung disease (ILD) with a progressive phenotype, except Idiopathic pulmonary fibrosis (IPF)
* Initiation of nintedanib as first antifibrotic therapy according to physician´s decision which has been made as part of routine care prior to and independent of study inclusion
* Outpatients not currently hospitalized with a life expectancy > 12 months per investigator's assessment
* Written informed consent prior to study participation
* Current Forced vital capacity (FVC) measurement (taken within the last 3 months) available in the patient file
* Women of childbearing potential must take appropriate precautions against getting pregnant during the intake of nintedanib.

Exclusion Criteria:

* Patients with contraindications according to Summary of product characteristics (SmPC)
* Prior use of any antifibrotic treatment
* Lack of informed consent
* Pregnant or lactating females
* Any physician diagnosed exacerbation of Interstitial lung disease (ILD) in the patient's history file, irrespective of time since event
* Current diagnosis of lung cancer
* Respiratory failure (pH < 7,35 and/ or respiratory rate > 30/min) in the patient's history
* Participation in a parallel interventional clinical trial
* Patients being spouse or lateral relatives to the second degree or economically dependent from the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic fibrosing Interstitial lung disease (ILD) with a progressive phenotype excluding Idiopathic Pulmonary Fibrosis (IPF) patients.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Correlation between change from baseline to week 52 in Forced vital capacity (FVC) [% pred.] and change from baseline to week 52 in dyspnea symptom score | Up to week 52
  The "living with pulmonary fibrosis" (L-PF) questionnaire for dyspnea/cough symptom score consists of 44 items divided into two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module assesses shortness of breath (dyspnea), cough and fatigue over the last 24 hours. The Impacts module assesses multiple aspects of health related quality of life (HRQoL) over the last 7 days. Symptoms and Impacts scores are used to calculate a total score.
  •Items in both modules have response options on a five-option numeric rating score with an anchor of 0 "Not at all" to 4 "Extremely". Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
Correlation between change from baseline to week 52 in Forced vital capacity (FVC) [% pred.] and change from baseline to week 52 in cough symptom score | Up to week 52
  The "living with pulmonary fibrosis" (L-PF) questionnaire for dyspnea/cough symptom score consists of 44 items divided into two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module assesses shortness of breath (dyspnea), cough and fatigue over the last 24 hours. The Impacts module assesses multiple aspects of HRQoL over the last 7 days. Symptoms and Impacts scores are used to calculate a total score.
  •Items in both modules have response options on a five-option numeric rating score with an anchor of 0 "Not at all" to 4 "Extremely". Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.

SECONDARY OUTCOMES:
Correlation between change from baseline to week 52 in Forced vital capacity (FVC) [millilitres mL] and change from baseline to week 52 in dyspnea symptom score | Up to week 52
  The "living with pulmonary fibrosis" (L-PF) questionnaire for dyspnea/cough symptom score consists of 44 items divided into two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module assesses shortness of breath (dyspnea), cough and fatigue over the last 24 hours. The Impacts module assesses multiple aspects of HRQoL over the last 7 days. Symptoms and Impacts scores are used to calculate a total score.
  •Items in both modules have response options on a five-option numeric rating score with an anchor of 0 "Not at all" to 4 "Extremely". Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
Correlation between change from baseline to week 52 in Forced vital capacity (FVC) [millilitres mL] and change from baseline to week 52 in cough symptom score | Up to week 52
  The "living with pulmonary fibrosis" (L-PF) questionnaire for dyspnea/cough symptom score consists of 44 items divided into two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module assesses shortness of breath (dyspnea), cough and fatigue over the last 24 hours. The Impacts module assesses multiple aspects of HRQoL over the last 7 days. Symptoms and Impacts scores are used to calculate a total score.
  •Items in both modules have response options on a five-option numeric rating score with an anchor of 0 "Not at all" to 4 "Extremely". Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
Absolute change from baseline in living with pulmonary fibrosis (L-PF) cough symptom score [points] at week 52 | At week 52
  The "living with pulmonary fibrosis" (L-PF) questionnaire for dyspnea/cough symptom score consists of 44 items divided into two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module assesses shortness of breath (dyspnea), cough and fatigue over the last 24 hours. The Impacts module assesses multiple aspects of HRQoL over the last 7 days. Symptoms and Impacts scores are used to calculate a total score.
  •Items in both modules have response options on a five-option numeric rating score with an anchor of 0 "Not at all" to 4 "Extremely". Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
Absolute change from baseline in living with pulmonary fibrosis (L-PF) dyspnea symptom score [points] at week 52 | At week 52
  The "living with pulmonary fibrosis" (L-PF) questionnaire for dyspnea/cough symptom score consists of 44 items divided into two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module assesses shortness of breath (dyspnea), cough and fatigue over the last 24 hours. The Impacts module assesses multiple aspects of HRQoL over the last 7 days. Symptoms and Impacts scores are used to calculate a total score.
  •Items in both modules have response options on a five-option numeric rating score with an anchor of 0 "Not at all" to 4 "Extremely". Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.

CONTACTS AND LOCATIONS:
Locations (30):
- Bulgaria (2):
  - Acibadem City Clinic Tokuda University Hospital EAD, Sofia
  - Medical Military Academy MHAT Sofia, Sofia
- Czechia (5):
  - University Hospital Brno, Brno
  - Nemocnice AGEL Novy Jicin a.s., Nový Jičín
  - University Hospital Ostrava, Ostrava-Poruba
  - Fakultni Nemocnice Plzen, Pilsen
  - Thomayer University Hospital, Prague
- Poland (8):
  - Szpital Uniwersytecki Nr 2 Im Dr Jana Biziela W Bydgoszczy, Bydgoszcz
  - Mirosław Nęcki SPL, Krakow
  - Somed Cr Sp. z o.o. sp.k., Lodz
  - IPL Michał Krawczyk, Lodz
  - Indywidualna SPL Małgorzata Noceń-Piskorowska, Szczecin
  - Biomedical Centers Sp. z o.o., Warsaw
  - Prywatna Praktyka Lekarska Paweł Piesiak, Wroclaw
  - Hanna Jagielska Len IPL, Zielona Góra
- Romania (12):
  - Dr. Ion Cantacuzino Clinical Hospital, Bucharest
  - Strambu I. Irina-Ruxandra - Activitate Medicala, Bucharest
  - Dr. Belaconi I. Ionela-Nicoleta - Medic Specialist Pneumologie, Bucharest
  - Dr. Toma Claudia Lucia - Medic Primar Pneumologie, Bucharest
  - Bronz Media SRL, Cluj-Napoca
  - Doctor 4 Sim Srl, Cluj-Napoca
  - PFI Ramazan Ana-Maria, Constanța
  - Sc Pneumo Clinic Dantes Srl, Constanța
  - Pneumo Research Srl, Moşniţa Nouă
  - Spital De Pneumologie Dr. Lavinia Davidescu S.R.L., Oradea
  - Dr. Fira-Mladinescu SRL, Timișoara
  - Iasis Srl, Timișoara
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - HOCH Health Ostschweiz, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com